CLINICAL TRIAL: NCT00707317
Title: Prospective Head-to-head Comparison of the Two Commercially Available Approved TIGRA (QuantiFERON-TB Gold In-Tube and T.SPOT.TB) With the Established Mendel-Mantoux Skin-test in Immunocompromized Patients
Brief Title: T Cell Interferon-gamma Release Assay (TIGRA) in Immunocompromised Individuals
Acronym: TBNET-TIPS
Status: Completed | Type: Observational
Sponsor: Tuberculosis Network European Trialsgroup (Network)
Responsible Party: Principal Investigator, Martina Sester, PhD, Professor, Tuberculosis Network European Trialsgroup
Other Study IDs: TBNET-TIGRA
Record Dates: First submitted 2008-06-25; First posted 2008-06-30 (Estimated); Last update posted 2015-12-16 (Estimated); Status verified 2015-12

CONDITIONS: Tuberculosis; Monitoring, Immunologic
Keywords: M. tuberculosis; latent tuberculosis infection; Quantiferon assay; ELISPOT assay; tuberculin skin test; immunocompromised patients
MeSH Terms: conditions — Tuberculosis; Latent Tuberculosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma supernatants of stimulated samples for cytokine analysis.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (7):
- 1: HIV infected individuals
- 2: patients with chronic renal failure
- 3: patients after solid organ transplantation (lung, liver, kidney, kidney-pancreas)
- 4: patients with rheumatoid arthritis
- 5: stem cell transplant recipients
- 6: immunocompromised patients with confirmed tuberculosis
- 7: immunocompetent controls with no known risk of exposure or tuberculosis

SUMMARY:
Until recently, the tuberculin skin test (TST) was the only available diagnostic assay for detection of latent infection with M. tuberculosis (LTBI). Despite the low overall incidence of symptomatic tuberculosis infection in low-prevalence countries, the potential mortality and morbidity mandate constant vigilance to identify patients at risk for reactivation. Due to systemic immunosuppression, immunocompromised patients with latent M. tuberculosis infection are at increased risk of progression to active disease. This applies to patients with various causes of immunodeficiency such as HIV-infected patients, allogeneic stem cell and solid organ transplant recipients, patients with rheumatoid arthritis and patients with chronic renal failure. Therefore, current guidelines aimed at preventing tuberculosis infection in immunocompromized individuals recommend a generalized screening for evidence of latent infection to target appropriate preventative prophylaxis. At present, tuberculosis control programs exclusively rely on the tuberculin skin test to identify a latent infection in asymptomatic individuals.

Recently, novel in vitro assays termed T cell interferon-gamma release assay (TIGRA) have become available that are based on the detection of interferon-gamma (IFN-gamma) production in T cells or supernatants after stimulation with highly specific antigens of M. tuberculosis. Two TIGRA are commercially available, the ELISPOT based T.SPOT.TB and the ELISA based QuantiFERON-TB Gold test (now available as an "IN-TUBE" version).

The aim of the study is a prospective comparison of the two commercially available approved TIGRA (QuantiFERON-TB Gold In-Tube and T.SPOT.TB) with the established Mendel-Mantoux skin-test in immunocompromized patients (main focus on sensitivity and specificity).

The study hypotheses are as follows:

1. In immunocompromised patients, the two commercially available approved TIGRA (QuantiFERON-TB Gold In-Tube and T.SPOT.TB) have increased sensitivity and specificity as compared to the established Mendel-Mantoux skin-test.
2. Results from QuantiFERON-TB Gold In-Tube and T.SPOT.TB do not differ in immunocompromised patients.

DETAILED DESCRIPTION:
Until recently, the tuberculin skin test (TST) was the only available diagnostic assay for detection of latent infection with M. tuberculosis (LTBI). Despite the low overall incidence of symptomatic tuberculosis infection in low-prevalence countries, the potential mortality and morbidity mandate constant vigilance to identify patients at risk for reactivation. Due to systemic immunosuppression, immunocompromised patients with latent M. tuberculosis infection are at increased risk of progression to active disease. This applies to patients with various causes of immunodeficiency such as HIV-infected patients, allogeneic stem cell and solid organ transplant recipients, patients with rheumatoid arthritis and patients with chronic renal failure. Therefore, current guidelines aimed at preventing tuberculosis infection in immunocompromized individuals recommend a generalized screening for evidence of latent infection to target appropriate preventative prophylaxis. At present, tuberculosis control programs exclusively rely on the tuberculin skin test to identify a latent infection in asymptomatic individuals.

Recently, novel in vitro assays termed T cell interferon-gamma release assay (TIGRA) have become available that are based on the detection of interferon-gamma (IFN-gamma) production in T cells or supernatants after stimulation with highly specific antigens of M. tuberculosis. Two TIGRA are commercially available, the ELISPOT based T.SPOT.TB and the ELISA based QuantiFERON-TB Gold test (now available as an "IN-TUBE" version). Current evidence suggests that TIGRA based on cocktails containing ESAT-6 and CFP-10 have the potential to become useful diagnostic tools. It has, however, been shown, that rates of indeterminate and positive results may differ between both tests, suggesting that they might provide different results in routine clinical practice. Moreover, there is only inadequate evidence on the value of those TIGRA in the management of immunocompromised individuals. Based on the current literature and most recent meta-analyses, there is an urgent need for head-to-head comparative studies of the two commercially available tests in immunocompromised patients. This study is designed to carry out a head-to-head comparison of the T.SPOT.TB and the ELISA based QuantiFERON-TB Gold In-Tube test with the TST in immunosuppressed populations. In a second step that will be addressed at a later stage, this study may be extended to longitudinally assess the predictive value of a positive blood test for progression to active disease.

The study will be performed within the tuberculosis network european trialsgroup (TBNET). It will be performed in a multicenter setting involving 23 participating centers from a total of 14 european countries. The study aims to include a total of 1800 study subjects distributed as follows: 200 HIV infected individuals with high and low CD4 T cells/µl (above and below 250 CD4 T cell/µl), respectively, 200 patients with chronic renal failure, 200 stem cell transplant recipients, 200 solid organ transplantation (lung, liver, kidney, kidney-pancreas) patients, 200 patients with rheumatoid arthritis. In addition, 200 immunocompromised patients with confirmed tuberculosis, 200 immunocompetent individuals with similar risk factors as patients, and 200 immunocompetent controls with no known risk of exposure or tuberculosis will serve as control groups.

ELIGIBILITY:
Inclusion Criteria:

* Individual as specified for the study population
* Written informed consent
* Indication to perform tuberculin skin test(suspect latent infection, according to standard guidelines, differential diagnosis)

Exclusion Criteria:

* <18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: immunocompetent and immunocompromised patients
Sampling Method: Non-Probability Sample
Enrollment: 1843 (Actual)
Dates: Start 2008-06; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
IGRA performance | at the time of analysis
  performance of two IGRAs and skin test in immunocompromised patients

SECONDARY OUTCOMES:
active tuberculosis on follow-up | variable follow-up on all patients
  Active TB on follow-up depending on test result

CONTACTS AND LOCATIONS:
Overall Officials: Martina Sester, PhD, Principal Investigator — Department of Transplant and Infection Immunology, University of the Saarland, 66421 Homburg; Christoph Lange, MD, PhD, Study Chair — Div. of Clinical Infectious Diseases, Medical Clinic, Research Center Borstel, Germany
Locations (21):
- Cellestis Limited, Carnegie, Australia
- National Center of Infectious and Parasitic Diseases, Sofia, Bulgaria
- Herlev Hospital, Herlev, Denmark
- Germany (4):
  - Research Center Borstel, Borstel
  - HIV Treatment and Clinical Research Unit, Frankfurt
  - Department of Infectious Diseases, Univ. of Freiburg, Freiburg im Breisgau
  - University of the Saarland, Homburg
- Respiratory Medicine, University of Thessaly, Mezourlo-Larissa, Greece
- Italy (3):
  - Emerging Bacterial Pathogens Unit, Milan
  - National Institute for Infectious Diseases L. Spallanzani, Roma
  - WHO Collaborating Center for TB and Lung Diseases, Tradate
- KNCV Tuberculosis Foundation, The Hague, Netherlands
- Centro de Diagnóstico Pneumológico, Lisbon, Portugal
- Clinica de Pneumologie, Marius Nasta Institute of Pneumology, Bucharest, Romania
- Servei de Microbiologia, Barcelona, Spain
- Karolinska Institute, Stockholm, Sweden
- Centre Antituberculeux, Hôpital Cantonal Universitarie, Geneva, Switzerland
- Turkey (Türkiye) (2):
  - Baþkent Üniversitesi Týp Fakültesi, Ankara
  - Department of Chest Diseases and Tuberculosis, Ankara
- United Kingdom (2):
  - Chest Clinic, London
  - Imperial College London, London

REFERENCES:
- [Result] Sester M, van Leth F, Bruchfeld J, Bumbacea D, Cirillo DM, Dilektasli AG, Dominguez J, Duarte R, Ernst M, Eyuboglu FO, Gerogianni I, Girardi E, Goletti D, Janssens JP, Julander I, Lange B, Latorre I, Losi M, Markova R, Matteelli A, Milburn H, Ravn P, Scholman T, Soccal PM, Straub M, Wagner D, Wolf T, Yalcin A, Lange C; TBNET. Risk assessment of tuberculosis in immunocompromised patients. A TBNET study. Am J Respir Crit Care Med. 2014 Nov 15;190(10):1168-76. doi: 10.1164/rccm.201405-0967OC. PMID 25303140
- [Result] Lange C, van Leth F, Sester M; TBnet. Viral Load and Risk of Tuberculosis in HIV Infection. J Acquir Immune Defic Syndr. 2016 Feb 1;71(2):e51-3. doi: 10.1097/QAI.0000000000000834. No abstract available. PMID 26761521
- See also: TBNET website — http://www.tb-net.org/